CLINICAL TRIAL: NCT05959031
Title: Exploring the Parameter Space of High Frequency Magnetic Perturbation in Manipulating Neural Excitability and Plasticity.
Brief Title: Parameter Space of kTMP
Acronym: SBIR_2022
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Magnetic Tides (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: MagneticTides
Record Dates: First submitted 2023-06-27; First posted 2023-07-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active kTMP (Experimental): Participants received 0.5 - 8 V/m of active stimulation.
  Interventions: Device: kTMP
- sham kTMP (Sham Comparator): Participants received 0.01 V/m of sham stimulation.
  Interventions: Device: Sham kTMP

INTERVENTIONS:
Device: kTMP — a new non-invasive brain stimulation tool
  Arms: active kTMP
Device: Sham kTMP — a new non-invasive brain stimulation tool with sham setting selected
  Arms: sham kTMP

SUMMARY:
The investigators have recently developed a new non-invasive brain stimulation (NIBS) system, kilohertz transcranial magnetic perturbation (kTMP) that opens up a new experimental space for safely modulating neural excitability in targeted areas of the human brain. This project will characterize the broad parameter space of kTMP in terms of tolerability and efficacy in healthy individuals. Following earlier feasibility studies, we are now increasing our number of subjects in order to capture preliminary safety and effectiveness information on a near-final device.

DETAILED DESCRIPTION:
Non-invasive brain stimulation (NIBS) has attracted considerable interest in the cognitive neuroscience community, providing an important basic research tool to study brain function, with emerging clinical applications to enhance function in individuals with neurological disorders.

The investigators have developed a radically new NIBS approach, one in which subthreshold modulation of neural excitability is brought about via oscillating magnetic fields at kilohertz (kHZ) frequencies. This system, referred to kTMP (kHz Transcranial Magnetic Perturbation) significantly increases the range of subthreshold E-field induction, and through modulation of the envelope of the kHz carrier frequency, can impose E-fields at physiological relevant frequencies. The investigators will conduct testing with healthy human participants to assess the tolerability and efficacy of the system in producing changes in cortical physiology.

ELIGIBILITY:
Inclusion Criteria:

Age 18-75

Exclusion Criteria:

* serious medical condition
* had a seizure of any sort
* epilepsy or experienced seizures
* neurological disorder
* head injury
* stroke
* had any form of brain surgery
* history of migraine
* metal implants in your head, excluding the mouth
* pacemaker
* implanted medical devices of any sort
* pregnant
* hearing loss or hearing impairments
* jet lag
* stress
* substance abuse
* highly stressful event over the past 24 hours
* broken or abnormal skin on your scalp

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported sensation/discomfort through questionnaire during kTMP stimulation. | Measures will be obtained 4-5 seconds after each kTMP stimulation at a specific E-field (when the visual display appears on the screen), in total 16 times throughout the kTMP stimulation trial.
  As per the FDA's guidance (www.fda.gov/media/81784/download) on device feasibility studies, initiation of an early feasibility study must be justified by an appropriate benefit-risk analysis and adequate human subject protection measures. This outcome measures device feasibility in terms of device tolerability. To estimate the stimulation threshold, the investigators will use an adaptive procedure in which they sequentially increase the stimulation intensity (E-field amplitude) and register self-reports of sensation. Stimulation intensity will start from 0.01 V/m (sham) increasing 0.5 V/m at a time for 16 trials until it reaches 7.6 V/m. Participants provided three ratings using an 11-point scale (0 = not at all; 10 = extremely) in response to questions on annoyance, pain, and muscle twitching. ("How annoying was kTMP?", "How painful was kTMP?", and "If there were any muscle twitches from the kTMP, how strong were they?") A higher score means more sensation/discomfort.
Self-reported sensation/discomfort through questionnaire after kTMP stimulation. | Measures will be obtained 1 minute after kTMP stimulation.
  As per the FDA's guidance (www.fda.gov/media/81784/download) on device feasibility studies, initiation of an early feasibility study must be justified by an appropriate benefit-risk analysis and adequate human subject protection measures. This outcome measures device feasibility in terms of device tolerability. After the kTMP stimulation, the investigators will register self-reports of sensation from the participant to see any lasting effect in terms of sensation. Participants provided three ratings using an 11-point scale (0 = not at all; 10 = extremely) in response to questions on annoyance, pain, and muscle twitching. ("How annoying was kTMP?", "How painful was kTMP?", and "If there were any muscle twitches from the kTMP, how strong were they?") A higher score means more sensation/discomfort.
Motor evoked potential (MEPs) amplitude recorded with electromyography (EMG) before kTMP stimulation. | Measures will be obtained from 0 to 15 minutes before the stimulation.
  This outcome measures device feasibility in terms of efficacy, as MEP changes indicate changes in cortical excitability induced by kTMP. As an operational definition of cortical excitability, the investigators will measure MEPs recorded in a peripheral hand muscle through the EMG system. The threshold procedure will be first conducted using single-pulse Transcranial magnetic stimulation (TMS) to find the M1 hotspot and threshold intensity. Once the threshold is set, MEPs will be obtained using the single-pulse and paired-pulse TMS procedures. These measurements will be taken prior to the experimental intervention of kTMP to obtain a baseline measure.
Motor evoked potential (MEPs) amplitude recorded with EMG after kTMP stimulation. | Measures will be obtained 1 hour 30 minutes after the stimulation.
  This outcome measures device feasibility in terms of efficacy, as MEP changes indicate changes in cortical excitability induced by kTMP. After the kTMP stimulation as a plasticity-inducing technique, we obtain MEPs using the single-pulse and paired-pulse TMS procedures. MEPs will be recorded in a peripheral hand muscle through the EMG system. The primary intervention of interest is the kTMP system, with various manipulations of the parameter settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Magnetic Tides, El Cerrito, California, United States

IPD SHARING:
Plan to Share IPD: Undecided